CLINICAL TRIAL: NCT05278845
Title: A Phase 1, Open-Label, Randomized, Crossover Study to Evaluate the Effect of Food on the Pharmacokinetics of SLC-391 in Healthy Adult Subjects
Brief Title: Crossover Study to Evaluate the Effect of Food on the Pharmacokinetics of SLC-391 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SignalChem Lifesciences Corporation (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SLC-391-103
Record Dates: First submitted 2022-02-08; First posted 2022-03-14 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Food-drug Interaction

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in a 1:1 ratio to one of two treatment sequences with 11 subjects per treatment sequence as outlined below. Each subject will receive both treatments (Treatment A and Treatment B) with a washout period of at least 7 days between successive SLC-391 single doses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Sequence 1 (Experimental): SLC-391 10 mg capsules (manufactured by China Gateway Pharmaceutical Development Co. (Shanghai, P.R. China)) administered as 5 x 10 mg capsules under fasted conditions.
  Interventions: Drug: SLC-391
- Treatment Sequence 2 (Experimental): SLC SLC-391 10 mg capsules (manufactured by China Gateway Pharmaceutical Development Co. (Shanghai, P.R. China)) administered as 5 x 10 mg capsules under fed conditions.
  Interventions: Drug: SLC-391

INTERVENTIONS:
Drug: SLC-391 — SLC-391 is an AXL inhibitor

SUMMARY:
This will be a single center, Phase 1, open-label, randomized, single dose, 2-period, 2-sequence, crossover study to evaluate the PK, safety, and tolerability of a single oral dose of SLC-391 under fed and fasted conditions in approximately 22 healthy male and non-childbearing potential female subjects.

Subjects will be randomized in a 1:1 ratio to one of two treatment sequences with 11 subjects per treatment sequence. Each subject will receive both treatments (Treatment A and Treatment B) with a washout period of at least 7 days between successive SLC-391.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
2. Male or non-childbearing potential female, non-smoker (no use of tobacco or nicotine products within 3 months prior to screening, confirmed by cotinine test), ≥18 and ≤55 years of age, with body mass index (BMI) >18.5 and <30 kg/m2 and body weight ≥50.0 kg for males and ≥45.0 kg for females.
3. Healthy as defined by:

   1. The absence of clinically significant illness and/or surgery within 4 weeks prior to dosing.
   2. The absence of clinically significant history of neurological, endocrine, cardiovascular, respiratory, hematological, immunological, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease.
4. Non-childbearing potential female defined as:

   1. Post-menopausal (spontaneous amenorrhea for at least 12 months prior to dosing) with confirmation by documented follicle stimulating hormone (FSH) levels ≥ 40 mIU/mL; or
   2. Surgically sterile (bilateral oophorectomy, hysterectomy or tubal ligation at least 3 months prior to dosing, verified through medical records). If surgical sterility cannot be verified, female subjects who are sexually active with a non-sterile male partner (sterile male partners are defined as men vasectomized for at least 3 months prior to dosing) must be willing to use one of the following acceptable contraceptive methods throughout the study and for 90 days after the last dose:

   (i) Simultaneous use of hormonal contraceptive (e.g., oral, patch, depot injection, implant, vaginal ring, intrauterine device) or non-hormonal intrauterine device used for at least 4 weeks prior to dosing (must agree to use the same contraceptive throughout the study) and condom for the male partner; (ii) Simultaneous use of diaphragm or cervical cap with spermicide and condom for the male partner, started at least 21 days prior to dosing.
5. Male subjects who are sexually active with a female partner of childbearing potential (childbearing potential females are defined as women that are neither post-menopausal nor surgically sterile) must be willing to use one of the following acceptable contraceptive methods from the first dose and for 90 days after the last dose, unless they can provide medical records indicating that they have been vasectomized for at least 3 months prior to dosing:

   1. Simultaneous use of condom and, for the female partner, hormonal contraceptives used since at least 4 weeks prior to sexual intercourse or intrauterine contraceptive device placed for at least 4 weeks prior to sexual intercourse;
   2. Simultaneous use of condom with spermicide and a diaphragm or cervical cap for the female partner.
6. Male subjects must be willing not to donate sperm during the study and for 90 days after the last dose.
7. Willing and able to comply with all scheduled visits, treatment plan, laboratory tests and all other required study procedures.

Exclusion Criteria:

1. Any clinically significant abnormality at physical examination, clinically significant abnormal laboratory test results or positive test for human immunodeficiency virus (HIV) antigen, hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibody found during medical screening.
2. Positive urine drug screen, alcohol breath test or urine cotinine test at screening.
3. History of allergic reactions to SLC-391 or to any excipient in the formulation.
4. History of clinically significant allergy or hypersensitivity to any drug or food or other substance.
5. History of lactose or galactose intolerance, lactase deficiency, or glucose-galactose malabsorption.
6. Positive pregnancy test at screening or breastfeeding subject.
7. Male subjects with partners that are currently pregnant or planning to become pregnant during the study or within 30 days following the last dose of the study drug.
8. Clinically significant ECG abnormalities (Fridericia's corrected QT interval [QTcF] ≥450 msec) or vital sign abnormalities (systolic blood pressure [BP] lower than 90 or over 140 mmHg, diastolic BP lower than 50 or over 90 mmHg, heart rate [HR] less than 50 or over 100 beats per minute [bpm]), or respiratory rate (RR) less than 8 or over 20 respirations per minute (rpm) at screening.
9. History of or a family history of congenital QT prolongation or with a history of risk factors for torsade de pointes (e.g., heart failure, hypokalemia, family history of long QT Syndrome), or use of concomitant medications that prolong the QT/ QT interval corrected for HR (QTc interval).
10. History or presence of sustained or symptomatic bradycardia (≤40 bpm), left bundle branch block, ventricular arrhythmia excluding premature ventricular contractions (PVCs) or uncontrolled ventricular arrhythmia. Subjects with a supraventricular arrhythmia not requiring medical treatment and a normal ventricular rate are eligible.
11. History of alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to screening that exceeds 10 units for women or 15 units for men of alcohol per week (1 unit = 340 mL of beer 5%, 140 mL of wine 12%, or 45 mL of distilled alcohol 40%).
12. History of drug abuse within 1 year prior to screening or recreational use of soft drugs (such as marijuana) within 1 month or hard drugs (such as cocaine, phencyclidine [PCP], crack, opioid derivatives including heroin, and amphetamine derivatives) within 3 months prior to screening.
13. Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days prior to the first dose, administration of a biological product in the context of a clinical research study within 90 days prior to the first dose, or concomitant participation in an investigational study involving no drug or device administration.
14. Use of medications for the timeframes specified below, with the exception of medications exempted by the Investigator on a case-by-case basis because they are judged unlikely to affect the PK profile of the study drug or subject safety (e.g., topical drug products without significant systemic absorption):

    1. Prescription medications within 14 days prior to the first dose (except hormonal contraception);
    2. Any vaccination, including COVID-19 vaccine, within 14 days prior to the first dose or a live or live-attenuated vaccine within 30 days prior to the first dose;
    3. Over-the-counter products and natural health products (including herbal remedies, homeopathic and traditional medicines, probiotics, food supplements such as vitamins, minerals, amino acids, essential fatty acids, and protein supplements used in sports) within 7 days prior to the first dose, with the exception of the occasional use of acetaminophen (up to 2 g daily);
    4. Hormone replacement therapy within 28 days prior to the first dose of the study drug;
    5. Depot injection or implant of any drug within 3 months prior to the first dose;
    6. Any drugs known to induce or inhibit hepatic drug metabolism or renal clearance (e.g., erythromycin, cimetidine, barbiturates, phenothiazines, or herbal/plant derived preparations such as St. John's Wort, etc.) within 30 days prior to the first dose.
15. Donation of plasma within 7 days prior to first dosing. Donation or loss of blood (excluding volume drawn at screening) of 50 mL to 499 mL of blood within 30 days, or more than 499 mL within 56 days prior to the first dose.
16. Inability to swallow oral medication.
17. Presence of active gastrointestinal disease and/or other gastrointestinal conditions that interfere with motility, or are expected to interfere with the absorption, distribution, metabolism, or excretion of oral SLC-391.
18. Habitual consumption of more than 400 mg of caffeine per day.
19. Known or suspected active COVID-19 infection or contact with an individual with known COVID-19 within 14 days of screening.
20. A history or current evidence of any severe acute or chronic medical or psychiatric disorder or laboratory abnormality that might interfere with the subject's ability to provide informed consent, comply with the protocol or interfere with the interpretation of the study results.
21. Any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2022-02-12 (Actual); Primary Completion 2022-06-14 (Actual); Study Completion 2022-06-14 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of SLC-391 | 14 days
  Changes in AUC (AUC0-t and AUC0-inf) over time in subjects taking SLC-391 capsules administered as a single oral 50 mg dose under fasted and fed conditions in healthy adult subjects.
Maximum Observed Plasma Concentration (Cmax) | 14 days
  Cmax is the maximum observed plasma concentration in ng/mL

SECONDARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events (TEAEs) as assessed by NCI-CTCAE v5.0 | 35 days
  To assess TEAEs as criteria of safety of oral SLC-391
Number of Participants with Serious Adverse Events (SAEs) as assessed by NCI-CTCAE v5.0 | 35 days
  To assess SAEs as criteria of safety of oral SLC-391
Pharmacokinetic (PK) parameters calculated for SLC-391 in plasma concentrations: Tmax. | 14 days
  Tmax is the time in hours to reach Cmax following dosing.
Pharmacokinetic (PK) parameters calculated for SLC-391 in plasma concentrations: T½ el. | 14 days
  T½ el is the time in hours required for the plasma level of the study drug to decrease by one-half during the terminal elimination phase.
Pharmacokinetic (PK) parameters calculated for SLC-391 in plasma concentrations: Kel. | 14 days
  Kel is the elimination rate constant describing removal of the drug by all elimination processes including excretion and metabolism.
Pharmacokinetic (PK) parameters calculated for SLC-391 in plasma concentrations: Vd/F. | 14 days
  Vd/F is the apparent volume of distribution.
Pharmacokinetic (PK) parameters calculated for SLC-391 in plasma concentrations: Cl/F. | 14 days
  Cl/F is the apparent clearance.
Pharmacokinetic (PK) parameters calculated for SLC-391 in plasma concentrations: MRT. | 14 days
  MRT is the mean residence time.
Number of Participants with Clinically Significant Changes From Baseline in Laboratory Parameters | 14 days
  Laboratory investigation includes hematology, biochemistry, urinalysis, and Serology.
Number of Participants with Clinically Significant Changes From Baseline in Vital Signs | 14 days
  Vital sign measurements includes blood pressure, heart rate, respiratory temperature, and oral temperature.
Number of Participants with Clinically Significant Changes From Baseline in electrocardiogram (ECGs) Findings | 14 days
  ECG parameters includes heart rate, PR interval, QRS, QT, and QTcF.
Number of Participants with Clinically Significant Changes From Baseline in physical examinations | 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- Syneos Health Clinique Inc. (Quebec), Québec, Canada

IPD SHARING:
Plan to Share IPD: No